CLINICAL TRIAL: NCT04529772
Title: Phase 3, Randomized, Double-Blind, Placebo-Controlled Study of Acalabrutinib in Combination With Rituximab, Cyclophosphamide, Doxorubicin, Vincristine, and Prednisone (R-CHOP) in Subjects ≤75 Years With Previously Untreated Non-GCB DLBCL
Brief Title: A Combination of Acalabrutinib With R-CHOP in Subjects With Previously Untreated Non-GCB DLBCL (ACE-LY-312)
Acronym: ESCALADE
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Acerta Pharma BV (Industry)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D8227C00001; 2019-001755-39 (EudraCT Number)
Record Dates: First submitted 2020-08-25; First posted 2020-08-28 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Diffuse Large B-Cell Lymphoma
Keywords: Untreated Non-Germinal Center Diffuse Large B-Cell Lymphoma; Lymphoma; Lymphoma, B-Cell; Lymphoma, Large B-Cell, Diffuse; Neoplasms; Lymphoproliferative Disorders; Lymphatic Diseases; Lymphoma, Non-Hodgkin; Prednisone; Cyclophosphamide; Rituximab; Doxorubicin; Vincristine; Acalabrutinib; Calquence
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma; Lymphoma, B-Cell; Neoplasms; Lymphoproliferative Disorders; Lymphatic Diseases; Lymphoma, Non-Hodgkin | interventions — acalabrutinib; Prednisone; Rituximab; Cyclophosphamide; Vincristine; Doxorubicin

STUDY DESIGN:
Intervention Model Description: Double-blind Randomised Placebo-controlled Study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participant Care provider Investigator Outcomes assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- acalabrutinib + R-CHOP (Experimental): Acalabrutinib plus Rituximab, Cyclosphosphamide, Doxorubicin, Vincristine and Prednisone (R-CHOP)
  Interventions: Drug: acalabrutinib; Drug: Prednisone; Drug: Rituximab; Drug: Cyclophosphamide; Drug: Vincristine; Drug: Doxorubicin
- placebo + R-CHOP (Placebo Comparator): Placebo plus Rituximab, Cyclophosphamide, Doxorubicin, Vincristine and Prednisone (R-CHOP)
  Interventions: Drug: placebo; Drug: Prednisone; Drug: Rituximab; Drug: Cyclophosphamide; Drug: Vincristine; Drug: Doxorubicin

INTERVENTIONS:
Drug: acalabrutinib — Investigational Product
  Arms: acalabrutinib + R-CHOP
Drug: placebo — Placebo comparator
  Arms: placebo + R-CHOP
Drug: Prednisone — Investigational Product
Drug: Rituximab — Investigational Product
Drug: Cyclophosphamide — Investigational Product
Drug: Vincristine — Investigational Product
Drug: Doxorubicin — Investigational Product

SUMMARY:
Phase 3 randomized, double-blind, placebo-controlled, study assessing the efficacy and safety of acalabrutinib plus rituximab,cyclophosphamide, doxorubicin, vincristine, and prednisone (R-CHOP) vs placebo plus R-CHOP in subjects ≤75 years of age with previously untreated non-germinal center diffuse large B-cell lymphoma.

DETAILED DESCRIPTION:
Phase 3 randomized, double-blind, placebo-controlled, study to evaluate the efficacy and safety of acalabrutinib plus rituximab,cyclophosphamide, doxorubicin, vincristine, and prednisone (R-CHOP) as compared with placebo plus R-CHOP in subjects ≤75 years of age with previously untreated non-germinal center diffuse large B-cell lymphoma (activated B-cell (ABC) and unclassified).

ELIGIBILITY:
Inclusion Criteria:

* Men and women, age ≥18 and ≤75 years
* Pathologically confirmed DLBCL, sufficient diagnostic material should be available to forward to a central laboratory for gene expression profiling and pathology review.
* No prior treatment for DLBCL
* Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2.
* International Prognostic Index (IPI) score of 1 to 5
* Disease Stage II to IV by the Ann Arbor Classification
* Adequate organ and marrow function
* Agreement to use highly effective forms of contraception during the study and 12 months after the last dose of rituximab

Exclusion Criteria:

* Evidence of severe or uncontrolled systemic diseases
* Known history of a bleeding diathesis (i.e., haemophilia, von Willebrand disease)
* History of stroke or intracranial haemorrhage in preceding 6 months.
* Known CNS lymphoma or leptomeningeal disease
* Known primary mediastinal lymphoma
* Known High-grade B-cell lymphoma with MYC and BCL2 and/or BCL6 rearrangements
* Prior history of indolent lymphoma or CLL
* History of or ongoing confirmed PML
* Significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of first dose of study drug, or any Class 3 or 4 cardiac disease as defined by the New York Heart Association Functional Classification
* Malabsorption syndrome, disease significantly affecting gastrointestinal function, resection of the stomach, extensive small bowel resection that is likely to affect absorption, symptomatic inflammatory bowel disease, partial or complete bowel obstruction, or gastric restrictions and bariatric surgery, such as gastric bypass.
* Uncontrolled active systemic fungal, bacterial, viral, or other infection
* Prior anthracycline use ≥150 mg/m2

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 611 (Actual)
Dates: Start 2020-10-08 (Actual); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) per the Lugano Classification for NHL in Arm A compared to Arm B | at every single visit up to 60 months

SECONDARY OUTCOMES:
Investigator-assessed event-free survival (EFS) for NHL in Arm A compared to Arm B | at every single visit up to 60 months
Overall survival in Arm A compared to Arm B | at every single visit up to 60 months
Percentage of Participants Who Achieved a Complete Response (CR) per 2014 Lugano Classification for NHL | at every single visit up to 60 months

CONTACTS AND LOCATIONS:
Locations (206):
- United States (31):
  - Research Site, Tucson, Arizona
  - Research Site, Little Rock, Arkansas
  - Research Site, Irvine, California
  - Research Site, Aurora, Colorado
  - Research Site, Norwich, Connecticut
  - Research Site, Fort Myers, Florida
  - Research Site, Orlando, Florida
  - Research Site, St. Petersburg, Florida
  - Research Site, Tallahassee, Florida
  - Research Site, West Palm Beach, Florida
  - Research Site, Fort Wayne, Indiana
  - Research Site, Des Moines, Iowa
  - Research Site, Wichita, Kansas
  - Research Site, Louisville, Kentucky
  - Research Site, Baltimore, Maryland
  - Research Site, Grand Rapids, Michigan
  - Research Site, Minneapolis, Minnesota
  - Research Site, St Louis, Missouri
  - Research Site, Albany, New York
  - Research Site, New York, New York
  - Research Site, Stony Brook, New York
  - Research Site, Charlotte, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Eugene, Oregon
  - Research Site, Portland, Oregon
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Nashville, Tennessee
  - Research Site, Fort Sam Houston, Texas
  - Research Site, Lubbock, Texas
  - Research Site, Salem, Virginia
- Australia (10):
  - Research Site, Adelaide
  - Research Site, Camperdown
  - Research Site, Clayton
  - Research Site, Darlinghurst
  - Research Site, Heidelberg
  - Research Site, Hobart
  - Research Site, Kogarah
  - Research Site, Liverpool
  - Research Site, Nedlands
  - Research Site, Westmead
- Austria (3):
  - Research Site, Linz
  - Research Site, Salzburg
  - Research Site, Wels
- Belgium (3):
  - Research Site, Antwerp
  - Research Site, Bruges
  - Research Site, La Louvière
- Brazil (8):
  - Research Site, Curitiba
  - Research Site, Florianópolis
  - Research Site, Goiânia
  - Research Site, Passo Fundo
  - Research Site, Porto Alegre
  - Research Site, Ribeirão Preto
  - Research Site, Rio de Janeiro
  - Research Site, São Paulo
- Canada (9):
  - Research Site, Vancouver, British Columbia
  - Research Site, Toronto, CA
  - Research Site, Winnipeg, Manitoba
  - Research Site, London, Ontario
  - Research Site, Lévis, Quebec
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
  - Research Site, Ottawa
  - Research Site, Toronto
- China (18):
  - Research Site, Beijing
  - Research Site, Changchun
  - Research Site, Chengdu
  - Research Site, Guangzhou
  - Research Site, Hangzhou
  - Research Site, Harbin
  - Research Site, Jinan
  - Research Site, Luoyang
  - Research Site, Nanchang
  - Research Site, Nanning
  - Research Site, Shanghai
  - Research Site, Shenyang
  - Research Site, Shijiazhuang
  - Research Site, Suzhou
  - Research Site, Tianjin
  - Research Site, Wuhan
  - Research Site, Xiamen
  - Research Site, Zhengzhou
- Czechia (5):
  - Research Site, Brno
  - Research Site, Hradec Králové
  - Research Site, Ostrava - Poruba
  - Research Site, Pilsen
  - Research Site, Prague
- France (9):
  - Research Site, Brest
  - Research Site, Caen
  - Research Site, Marseille
  - Research Site, Montpellier
  - Research Site, Nantes
  - Research Site, Pessac
  - Research Site, Pierre-Bénite
  - Research Site, Rennes
  - Research Site, Toulouse
- Germany (5):
  - Research Site, Bamberg
  - Research Site, Berlin
  - Research Site, Dresden
  - Research Site, Homburg
  - Research Site, Neumünster
- India (6):
  - Research Site, Bangalore
  - Research Site, Delhi
  - Research Site, Kochi
  - Research Site, Mumbai
  - Research Site, Nashik
  - Research Site, Pune
- Israel (11):
  - Research Site, Afula
  - Research Site, Ashdod
  - Research Site, Beersheba
  - Research Site, Haifa
  - Research Site, Holon
  - Research Site, Jerusalem
  - Research Site, Nahariya
  - Research Site, Petah Tikva
  - Research Site, Ramat Gan
  - Research Site, Tel Aviv
  - Research Site, Ẕerifin
- Italy (18):
  - Research Site, Bari
  - Research Site, Bergamo
  - Research Site, Bologna
  - Research Site, Florence
  - Research Site, Genova
  - Research Site, Meldola
  - Research Site, Milan
  - Research Site, Novara
  - Research Site, Palermo
  - Research Site, Pavia
  - Research Site, Pisa
  - Research Site, Ravenna
  - Research Site, Reggio Emilia
  - Research Site, Roma
  - Research Site, Siena
  - Research Site, Torino
  - Research Site, Tricase
  - Research Site, Venezia
- Japan (20):
  - Research Site, Chiba
  - Research Site, Chūōku
  - Research Site, Fukuoka
  - Research Site, Itabashi-ku
  - Research Site, Kahoku-gun
  - Research Site, Kashiwa
  - Research Site, Kobe
  - Research Site, Kōtoku
  - Research Site, Kumamoto
  - Research Site, Kyoto
  - Research Site, Matsuyama
  - Research Site, Nagasaki
  - Research Site, Nagoya
  - Research Site, Niigata
  - Research Site, Okayama
  - Research Site, Osaka
  - Research Site, Sapporo
  - Research Site, Sendai
  - Research Site, Shimotsuke-shi
  - Research Site, Tsu
- Mexico (2):
  - Research Site, Chihuahua City
  - Research Site, Monterrey
- Poland (6):
  - Research Site, Gdansk
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Lublin
  - Research Site, Warsaw
  - Research Site, Wroclaw
- Portugal (5):
  - Research Site, Braga
  - Research Site, Lisbon
  - Research Site, Matosinhos Municipality
  - Research Site, Porto
  - Research Site, Vila Nova de Gaia
- Russia (3):
  - Research Site, Chelyabinsk
  - Research Site, Moscow
  - Research Site, Saint Petersburg
- South Korea (5):
  - Research Site, Busan
  - Research Site, Goyang-si
  - Research Site, Jeonju
  - Research Site, Seoul
  - Research Site, Suwon
- Spain (11):
  - Research Site, Alcalá de Henares
  - Research Site, Barcelona
  - Research Site, Gijón
  - Research Site, L'Hospitalet de Llobregat
  - Research Site, Madrid
  - Research Site, Palma
  - Research Site, Pamplona
  - Research Site, Pozuelo de Alarcón
  - Research Site, Salamanca
  - Research Site, Seville
  - Research Site, Valencia
- Taiwan (4):
  - Research Site, Kaohsiung City
  - Research Site, Tainan
  - Research Site, Taipei
  - Research Site, Taoyuan
- Turkey (Türkiye) (8):
  - Research Site, Ankara
  - Research Site, Balçova
  - Research Site, Edirne
  - Research Site, Izmir
  - Research Site, Kayseri
  - Research Site, Mersin
  - Research Site, Samsun
  - Research Site, Trabzon
- Ukraine (6):
  - Research Site, Cherkasy
  - Research Site, Khmelnytskyi
  - Research Site, Kyiv
  - Research Site, Lviv
  - Research Site, Mykolayiv
  - Research Site, Zaporizhzhia

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home